CLINICAL TRIAL: NCT00405548
Title: To Define in Human Preclinical Diastolic Dysfunction (PDD) the Actions of Chronic Administration of Subcutaneous (SQ) BNP on the Left Ventricular, Renal and Humoral Function and on the Integrated Response to Acute Sodium Loading
Brief Title: Human Brain Natriuretic Peptide (BNP) (or Nesiritide) to Help Heart, Kidney and Humoral Function.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Scios, Inc. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Horng Chen, Dr Horng H Chen, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 05-004190; P01HL076611 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Left Ventricular Diastolic Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BNP (nesiritide) (Active Comparator): BNP 10 micrograms/Kg twice per day given subcutaneously for 12 weeks
  Interventions: Drug: BNP (nesiritide)
- Placebo (Placebo Comparator): Saline solution given subcutaneously twice per day for 12 weeks (packaged to match active comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BNP (nesiritide)
  Other Names: natrecor; nesiritide
  Arms: BNP (nesiritide)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to evaluate the effects of cardiac hormone replacement with SQ (subcutaneous or under the skin) injection of BNP (brain natriuretic peptide, a hormone produced by the heart) on the pumping ability of the heart, kidney function and levels of different hormones in the blood in response to an intravenous salt solution.

DETAILED DESCRIPTION:
Prior to initiation of the study, subjects will be stabilized for at least one week on a no added salt diet (120 milliequivalent (mEq) Na/Day) which will be maintained during the study. Participants in this study will be randomized to receive BNP or placebo (an inactive, saline shot). The participant will need to give themselves a shot in their stomach (similar to diabetics giving themselves insulin) twice a day for twelve weeks. The study requires a screening visit to determine eligibility and discuss the study. At this visit a blood draw for heart and liver function and a six minute walk will be done. There will also be two other outpatient visits and two inpatient stays, for 48 hours, in the Clinical Research Unit at St. Marys Hospital. During the two overnight stays, blood and urine samples will be done to get heart and kidney function as well as a research echocardiogram. An acute saline load (0.9% normal saline 1.25 ml/kg/min for 1 hour) will be given and blood and urine samples collected After enrollment, the study lasts for twelve weeks. It is planned to treat 2 subjects with active drug per each placebo subject to improved the precision of between group comparison.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ejection fraction of greater than 50% with moderate or severe diastolic dysfunction as assessed by Doppler echocardiography
* No signs or symptoms of congestive heart failure and who have not been hospitalized for heart failure

Exclusion criteria:

* Myocardial Infarction (MI) within 3 months of screening
* Unstable angina within 14 days of screening, or any evidence of myocardial ischemia
* Significant valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
* Severe congenital heart diseases
* Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* Second or third degree heart block without a permanent cardiac pacemaker
* Stroke within 3 months of screening, or other evidence of significantly compromised central nervous system (CNS) perfusion
* Total bilirubin of > 1.5 mg/dL or other liver enzymes > 1.5 times the upper limit of normal (mg/dL = milligrams per deciliter)
* Serum creatinine of > 3.0 mg/dL
* Serum sodium of < 125 mEq/dL or > 160 mEq/dL (milliequivalents per deciliter)
* Serum potassium of < 3.5 mEq/dL or > 5.0/dL
* Serum digoxin level of > 2.0 ng/ml (nanograms per milliliter)
* Systolic pressure of < 85 mm Hg (millimeters of mercury)
* Hemoglobin < 10 gm/dl (grams per deciliter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-03; Primary Completion 2011-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horng H. Chen, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wan SH, McKie PM, Schirger JA, Slusser JP, Hodge DO, Redfield MM, Burnett JC Jr, Chen HH. Chronic Peptide Therapy With B-Type Natriuretic Peptide in Patients With Pre-Clinical Diastolic Dysfunction (Stage B Heart Failure). JACC Heart Fail. 2016 Jul;4(7):539-547. doi: 10.1016/j.jchf.2015.12.014. Epub 2016 Feb 10. PMID 26874387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 49 participants signed written informed consent to enroll in the study. Of these 8 were withdrawn prior to randomization for varying reasons.
Groups:
- BNP (Nesiritide): Brain Natriuretic Peptide (BNP) 10 micrograms/Kg twice per day given subcutaneously for 12 weeks
Period: Overall Study
Arm/Group | BNP (Nesiritide) | Placebo
Started | 28 | 13
Completed | 24 | 12
Not Completed | 4 | 1
Not completed — Cognitive Memory problems on study day | 1 | 0
Not completed — Amyloidosis on study echo-exclusionary | 0 | 1
Not completed — Unable to self-administer shots | 1 | 0
Not completed — Venous access failed during study day | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BNP (Nesiritide) | Placebo | Total
Number analyzed (Participants) | 24 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 17 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (8.1) | 69.6 (10.9) | 69.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 15 | 5 | 20
Region of Enrollment [Number; unit: participants]
  United States | 24 | 12 | 36

OUTCOME MEASURES:

1. Secondary Outcome: Change in Urinary Flow in Response to Saline Load
Description: Urinary flow is a measure of renal (or kidney) function and was measured in milliliters per minute.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | BNP (Nesiritide) | Placebo
Number analyzed (Participants) | 24 | 12
ml/minute | 4.2 (5.4) | -1.0 (2.1)
Statistical Analysis 1: Comparison: BNP (Nesiritide) vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Change in Glomerular Filtration Rate (GFR) in Response to Saline Load
Description: Renal or kidney function was measured by GFR determined by iothalamate clearance. GFR describes the flow rate of filtered fluid through the kidney measured in milliliters per minute per 1.73 m^2 of body surface area. A lower GFR means the kidney is not filtering normally. An estimated GFR of less than 60 mg/ml/1.73 m^2 of body surface area is considered to be impaired kidney function.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m^2 body surface area
Arm/Group | BNP (Nesiritide) | Placebo
Number analyzed (Participants) | 24 | 12
ml/min/1.73 m^2 body surface area | 6.8 (19.3) | 4.4 (27.3)
Statistical Analysis 1: Comparison: BNP (Nesiritide) vs Placebo; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

3. Primary Outcome: Change in Urinary Sodium Excretion in Response to Saline Load
Description: Renal (or kidney) function was measured by the sodium or salt in the urine, following administration of a pre-specified amount of saline (salt).
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: mEq/minute
Arm/Group | BNP (Nesiritide) | Placebo
Number analyzed (Participants) | 24 | 12
mEq/minute | 381.6 (450.8) | -10.5 (90.1)
Statistical Analysis 1: Comparison: BNP (Nesiritide) vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Left Ventricular (LV) Filling Pressure
Description: LV diastolic function as measured by Doppler echocardiography. E/e' is the ratio of the mitral inflow velocity (E) to the mitral annulus tissue Doppler velocity (e'). A decrease in the ratio indicates a lower filling pressure and improved LV diastolic function.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: E/e'
Arm/Group | BNP (Nesiritide) | Placebo
Number analyzed (Participants) | 24 | 12
E/e'
  Baseline LV Filling Pressure | 14.9 (4.1) | 14.9 (4.5)
  12 Week LV Filling Pressure | 12.6 (3.5) | 14.0 (5.1)
Statistical Analysis 1: Comparison: BNP (Nesiritide); Mean LV filling pressure was compared from baseline to 12 weeks within the BNP group; Test type: Superiority or Other; p = 0.004, t-test, 2 sided; A p-value of less 0.05 was considered to be statistically significant
Statistical Analysis 2: Comparison: Placebo; Mean LV filling pressure was compared from baseline to 12 weeks within the Placebo group; Test type: Superiority or Other; p = 0.43, t-test, 2 sided; A p-value of less 0.05 was considered to be statistically significant

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks during study with a 6 month follow-up telephone call to subject.
Arm/Group | BNP (Nesiritide) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 5/24 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNP (Nesiritide) (N=24) | Placebo (N=12)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heart Failure symptoms (Cardiac disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes